CLINICAL TRIAL: NCT05346887
Title: Home-based Early Intensive Hemiparesis Therapy: Engaging Nurture
Acronym: HEIGHTEN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-1981
Record Dates: First submitted 2022-03-28; First posted 2022-04-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy; Perinatal Stroke
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based Therapy (Experimental)
  Interventions: Behavioral: Home-based Therapy

INTERVENTIONS:
Behavioral: Home-based Therapy — The 18-week caregiver-delivered intervention involves daily 30-minute home-practice and weekly sessions with a therapist over video call or in-person at a local rehabilitation centre. During weekly sessions, the therapist will coach the caregiver(s), problem-solving with them and supporting their autonomy as agents of change in their child's care. The first 13-weeks of the program will be exclusively constraint-induced movement therapy, with bimanual therapy introduced in the last five weeks depending on child age. Intervention content will be individualized based on child age, ability, and interests.

SUMMARY:
The purpose of the study is to assess implementation and effectiveness of a caregiver-delivered rehabilitation intervention for infants and toddlers with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* aged three to 24 months (corrected, if premature)
* clinician-identified hand asymmetry
* suspected/confirmed cerebral palsy (hemiplegia or triplegia)
* willing to withhold other formal upper-limb focussed treatment during the study intervention - willing to commit to completing 18 weeks of daily home-practice and attending weekly therapy sessions.

Exclusion Criteria:

* participation in formal constraint induced movement therapy (CIMT) within last six months
* upper limb botulinum toxin A injections within previous six months
* brachial plexus injury
* lower motor neuron dysfunction
* upper limb congenital limb difference.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of therapists | <7 days after the 18-week intervention
  Satisfaction with the intervention will be assessed using a study-built questionnaire with Likert-scale response options 0 to 4, with 4 being greater satisfaction.
Canadian Occupational Performance Measure (COPM) | <7 days after the 18-week intervention
  Using the COPM, three to five individualized functional goals will be identified by caregivers and then scored on a scale of 1 to 10 for both Performance and Satisfaction.
Age-appropriate hand assessment (HAI/mini-AHA/AHA) | <7 days after the 18-week intervention
  The HAI/mini-AHA/AHA employ a video-recorded play-based session of <15 minutes to provide a logit-based measure of manual function.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 8 weeks +/-3days after the the 18-week intervention.
  Using the COPM, three to five individualized functional goals will be identified by caregivers and then scored on a scale of 1 to 10 for both Performance and Satisfaction.
Age-appropriate hand assessment (HAI/mini-AHA/AHA) | 8 weeks +/-3days after the the 18-week intervention.
  The HAI/mini-AHA/AHA employ a video-recorded play-based session of <15 minutes to provide a logit-based measure of manual function.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No